CLINICAL TRIAL: NCT03105817
Title: Study of Cellulose Triacetate Dialyzer (Solacea™): in Vivo Behavior in Hemodiafiltration-online
Brief Title: Cellulose Triacetate Dialyzer in Hemodiafiltration-online
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Infanta Leonor (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIB 09/2015
Record Dates: First submitted 2017-03-27; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-03

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: Asymmetric cellulose triacetate; Biocompatibility; Hemodiafiltration on-line; Convective volume; Adequacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Asymmetric cellulose triacetate (ATA™) — Each patient underwent 12 sessions of haemodialysis with the usual schedule, changing the usual dialyzer
  Other Names: Solacea™

SUMMARY:
In post-dilution haemodiafiltration only synthetic membranes have been used to date.

The allergy problems described with these membranes require the development of other membranes capable of performing this treatment. We describe in vivo performance and behaviour of an asymmetric cellulose triacetate(ATA™) membrane, to identify its depurative effectiveness and ease of use in clinical practice, as well as evaluate its biocompatibility in a single haemodialysis session (acute biocompatibility) and after one month of treatment (chronic).

DETAILED DESCRIPTION:
An interventional study was performed in 3 hemodialysis hospital units (La Princesa University Hospital, Príncipe de Asturias University Hospital and Infanta Leonor University Hospital, Community of Madrid, Spain) in which the usual dialyzer that each patient had for OLHDF was replaced with the Solacea™ dialyzer keeping the rest of the parameters unchanged. The study (LIB 09/2015) was reviewed and approved by the CEIC of the Príncipe de Asturias University Hospital.

* Design of the study Each patient underwent 12 sessions of haemodialysis with the usual schedule and monitor: 5008 of Fresenius (n=14), AK200US (n=5) and Artis of Gambro (n=3) and DBB007 of Nikkiso (n=1) all suitable for OLHDF, although with different convective transport control systems. The nursing staff connected the automatic OLHDF system. In the case where the system was Ultracontrol® (Gambro monitors) if alarm of PTM> 300 mmHg or system pressure (PSist)> 700 mmHg appeared and were not solved, Ultracontrol® would be withdrawn and the pressure-control system would be used.
* Data to be collected:

  1. Demographic and dialysis data

     * Demographic: sex, age, underlying disease, time in OLHDF, type of vascular access: fistula (AFV) and catheter (CT).
     * Dialysis Data: Monitor, dialysis fluid composition, sodium conductivity and bicarbonate concentration, dialysis fluid flow (Qd, ml min), liquid temperature, heparin type and dosage.
     * Each dialysis session: effective time (TE, min), blood flow (Qb, ml min), ultra-filtrated volume to achieve dry weight (UF, l/session), Vinf (l/session), infusion rate, (Qi, ml/min) Kt (l / session), maximum PTM and maximum Psist in Ultracontrol® (mmHg) and the technical complications, alarms and coagulation problems of the system that may appear.

     The filtration fraction (FF) was calculated as the percentage of Qi relative to Qb. The convective volume (Vconv) was defined as the total ultra-filtrated volume, which is the sum of VI and UF.7
  2. Analytical determinations

     1. Blood

        - On the first and last day of the study pre-dialysis samples were taken for the measurement of monocytes, IL-6 and IL-1β.
        * On the interval day of the first week, 3 blood samples were taken: 1st) at the beginning (CI), 2nd) at 30 min (CM) and the 3rd) at the end of the dialysis session (CP).

        In CI and CP the following parameters were measured: haemoglobin, proteins and albumin, urea, phosphorus, creatinine, uric acid, β2-microglobulin, myoglobin and retinol transport protein (RTP).

        Leukocytes, platelets, C3a and C5a were quantified in CI and CM.

        --- Laboratory determinations

        - General biochemical data: haemoglobin, proteins, albumin, urea, phosphorus, reactive protein C (PCR), creatinine and uric acid, β2-microglobulin, myoglobin, and (RTP) were determined with the usual analyser of each hospital.

        - Determinations of monocytes, complement, IL-6 and IL-1β were performed in the laboratory of the University of Alcalá:
        * Activation of plasma complement using a sandwich ELISA: Determination of C3a and C5a activation was performed on platelet rich plasma samples using commercially available ELISA kits C3a Elabscience (Wuhan, P.R. China) and ELISA C5a RayBiotech (Norcross, Georgia).
        * Determination of interleukin concentration in serum using a sandwich ELISA: IL-6 and IL-1β concentrations were measured in serum samples obtained from whole blood and stored at -80 ° C until use. Both kits used were supplied by Abcam (Cambridge, UK)
        * Determination of monocyte subpopulations: The different subpopulations of circulating monocytes in peripheral blood were identified by flow cytometry (FACSCalibur™, Becton Dickinson, San Jose, CA, USA). First of all, the monocyte population was selected according to size (FSC/forward scatter) and granularity (SSC/side scatter) and then the different subpopulations were selected by double immunofluorescence according to staining with the anti-CD14 conjugated Tricolor (monoclonal antibodies TuK4) and anti-CD16 conjugated FITC (monoclonal antibodies 3G8). Both antibodies and their respective isotype controls were purchased from Life Technologies Invitrogen (California, USA). The analysis was performed with the Cyflogic program.

          * Calculations The percentages of reduction (RR) were calculated with the formula: RR (%) = [(Cpre - Cpos) / Cpre] x 100, where Cpre and Cpos are the concentrations of the analysed substances pre- and post-dialysis.

        For protein bound substances and β2-microglobulin concentrations at the end of the session were corrected for haemoconcentration by a correction factor (FC) based on plasma protein concentration (PT):

        FC = PTpre / PTpos, where PTpre and PTpos are the total concentration of proteins pre-dialysis and post-dialysis.

        --- Statistical analysis All data was collected in a database (SPSS version 15). Each value was obtained with the average of the values obtained in the different sessions or analytical determinations.

        For the statistical analysis, descriptive tools were used, showing the average (standard deviation), median, quartiles or percentages as appropriate. For the comparison of two independent continuous variables, the Student t test for paired samples was used. For the comparison of more than two quantitative variables the ANOVA test was used. The p <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion

* Criteria:being over 18 years old, being treated with OLHDF for more than 4 weeks with 3 weekly sessions and sign an informed consent form.

Exclusion Criteria:

* pregnancy and illness that would make the patient's death predictable in less than 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-07-10 (Actual); Study Completion 2016-08-14 (Actual)

PRIMARY OUTCOMES:
Performance of asymmetric cellulose triacetate (ATA™) | One month
  Describing in vivo depurative efficacy of asymmetric cellulose triacetate (ATA™) measuring Kt, infusion volumen and clearance of RR of different molecules
Biocompatibility of asymmetric cellulose triacetate (ATA™) | One month
  Studying its acute (measuring complement and leukocites) and chronic (measuring monocytes subpopulationsand interleukines)
Clinical behaviour of ATA | One month
  Studuying alarm or clínical problemas related with dialyzer

CONTACTS AND LOCATIONS:
Locations (1):
- Marta Albalate Ramón, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maduell F, Navarro V, Hernandez-Jaras J, Calvo C. [Comparison of dialyzers in on-line hemodiafiltration]. Nefrologia. 2000 May-Jun;20(3):269-76. Spanish. PMID 10917004
- [Result] Sunohara T, Masuda T. Fundamental Characteristics of the Newly Developed ATA Membrane Dialyzer. Contrib Nephrol. 2017;189:215-221. doi: 10.1159/000451044. Epub 2016 Dec 12. PMID 27951571
- [Result] Sanchez-Villanueva RJ, Gonzalez E, Quirce S, Diaz R, Alvarez L, Menendez D, Rodriguez-Gayo L, Bajo MA, Selgas R. Hypersensitivity reactions to synthetic haemodialysis membranes. Nefrologia. 2014;34(4):520-5. doi: 10.3265/Nefrologia.pre2014.May.12552. English, Spanish. PMID 25036066
- [Result] Mineshima M. Optimal Design of Dialyzers. Contrib Nephrol. 2017;189:204-209. doi: 10.1159/000450802. Epub 2016 Dec 12. PMID 27951569
- [Result] Sunohara T, Masuda T. Cellulose triacetate as a high-performance membrane. Contrib Nephrol. 2011;173:156-163. doi: 10.1159/000329055. Epub 2011 Aug 8. PMID 21865788